CLINICAL TRIAL: NCT00190528
Title: Phase III Trial of Neoadjuvant Chemotherapy Followed by Surgery Versus Surgery Alone for Bulky Stage I/II Cervical Cancer: Japan Clinical Oncology Group Trial (JCOG0102)
Brief Title: A Trial of Neoadjuvant Chemotherapy + Surgery vs. Surgery for Bulky Stage I/II Cervical Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JCOG0102; C000000194
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Cervical Neoplasms
Keywords: cervical cancer; drug therapy; cisplatin; bleomycin; mitomycin; vincristine
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Neoadjuvant Therapy

ARMS (2):
- Surgery (Active Comparator)
  Interventions: Procedure: radical hysterectomy
- Chemotherapy + Surgery (Experimental)
  Interventions: Drug: neoadjuvant chemotherapy + radical hysterectomy

INTERVENTIONS:
Drug: neoadjuvant chemotherapy + radical hysterectomy
  Arms: Chemotherapy + Surgery
Procedure: radical hysterectomy
  Arms: Surgery

SUMMARY:
To investigate the clinical benefits of neoadjuvant chemotherapy for bulky stage I/II cervical cancer

DETAILED DESCRIPTION:
We designed this randomized study to investigate the clinical benefits of neoadjuvant chemotherapy for bulky stage I/II cervical cancer. Patients with FIGO stage I/II with bulky disease are randomized to either neoadjuvant chemotherapy (BOMP: Cisplatin 14mg/m2 day 1-5, Bleomycin 7mg day 1-5, Mitomycin 7mg/m2 day 5, and Vincristine 0.7mg/m2 day every 21 days for 2-4 cycles followed by radical hysterectomy or radical hysterectomy alone. The primary endpoint is overall survival and the secondary endpoints are progression-free survival, complication of surgery, completeness of radical hysterectomy, omission of postsurgical irradiation, completeness of postsurgical irradiation, response rate, and adverse events. A total 200 patients (100 per treatment arm) planned to accrue for this study within 5.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated cervical cancer
2. Pathologically diagnosed squamous carcinoma
3. FIGO stage Ib2, IIa (>4cm), and IIb
4. Measurable lesions
5. Possible to radical hysterectomy
6. Age: 20 to 70 years
7. PS: 0 and 1
8. WBC > 3,000/mm3, Hb > 9.0g/dl, Platelet > 100,000 /mm3, SGOT/SGPT < 60 IU/L, T-Bil < 1.5 mg/dL, Cr < 1.2 mg/dL, PaO2 > 80 torr, normal ECG
9. Written informed consent

Exclusion Criteria:

1. Patients who have any evidence of the other cancer present within the last 5 years with the exception of carcinoma in situ or intramucosal cancer those are curable with local therapy
2. Women during pregnancy or breast-feeding
3. Patients with psychiatric illness
4. Patients who have active infection
5. Patients who have uncontrolled diabetes or uncontrolled hypertension
6. Patients who have positive HBs
7. Patients who have had heart failure, unstable angina, or myocardial infarction within the past 6 months
8. Patients with interstitial pneumonitis or pulmonary fibrosis
9. Patients who are unable to undergo radical hysterectomy for complication of excessive obesity, liver cirrhosis, or bleeding tendency

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2002-02; Primary Completion 2004-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
progression-free survival
complication of surgery
completeness of radical hysterectomy
omission of postsurgical irradiation
completeness of postsurgical irradiation
response rate
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Toshiharu Kamura, MD, PhD, Study Chair — Kurume University
Locations (1):
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan

REFERENCES:
- See also: Related Info — http://www.jcog.jp/